CLINICAL TRIAL: NCT05612191
Title: An Open Label Post-Trial Access (PTA) of Catequentinib (AL3818, Anlotinib) Hydrochloride Mono or in Combination Therapies in Patients Who Have Completed an Advenchen Sponsored Oncology Study With AL3818 (A Compassionate Use Trial)
Brief Title: Catequentinib in Patients Who Have Completed an Advenchen Study (A Compassionate Use Trial)
Status: Available | Type: Expanded Access
Sponsor: Advenchen Laboratories, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AL3818-PTA
Record Dates: First submitted 2022-11-04; First posted 2022-11-10 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Sarcoma,Soft Tissue; Gynecologic Cancer
MeSH Terms: conditions — Sarcoma | interventions — anlotinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: AL3818 — It inhibits VEGFR2-mediated downstream signal transduction, thereby inhibiting tumor angiogenesis. It also has high potency against FGFr as well as VEGFr, and as such acts as a mainly dual inhibitor.
  Other Names: Catequentinib (AL3818, Anlotinib) Hydrochloride

SUMMARY:
Catequentinib (AL3818, Anlotinib) has been developed in a variety of clinical studies as single agents or in combination with others. This trial is designed to offer patients who completed an Advenchen sponsored AL3818 related study without progression the opportunity to continue to receive this investigational product in this Post-Trial Access study (a compassionate use trial), if the Investigator believes the patients can benefit from such a treatment and the patients have signed the Informed Consent Form.

DETAILED DESCRIPTION:
This is an open label trial and is designed to offer patients who are in a completed Advenchen sponsored AL3818 study without progression the opportunity to continue to receive AL3818. Qualified patients will continue therapy on their regimen established in the approved parent AL3818 clinical study until disease progression, physician decision, patient withdrawal, or sponsor discontinuation of the study. Dose modifications will be based on the suggestions in the approved parent AL3818 clinical study. Patients may be required to come to the site to receive AL3818. For patients who cannot come to the site to receive AL3818, the Site may mail the drug to the patient. The exact dispersing methods will be based on the Investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be currently receiving treatment with AL3818 on a previously approved parent protocol, including drug crossover patients.
* Patients must have achieved stable disease, partial response or complete response based on the most recent tumor assessment. If progressive disease on the most recent tumor assessment, the Investigator believes the patient can clinically benefit from continuing to receive AL3818.
* Female patients of child-bearing potential, and male partners must consent to use a medically acceptable method of contraception throughout the study period and for 4 months after the last dose of either study drug.
* Patient is willing and able to sign a new informed consent.
* Patients for whom the Investigator believes can benefit from continuing to receive AL3818

Exclusion Criteria:

* Patient has been discontinued from their previous AL3818 trial treatment greater than 3 weeks (one cycle) prior to entering the compassionate use trial.
* Patient progressed while receiving therapy with AL3818 during their participation in their immediate previous trial unless the Investigator believes the patient can clinically benefit from continuing to receive AL3818.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult